CLINICAL TRIAL: NCT00002998
Title: Phase II Study of Gemcitabine (GEMZAR) and Cisplatin (CDDP) in Advanced Breast Cancer
Brief Title: Gemcitabine and Cisplatin in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-963251; CDR0000065548 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + cisplatin (Experimental): Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 1 hour on days 1, 8, and 15 every 28 days. Patients with complete response may receive an additional 2 courses after attainment of complete response status. Treatment continues in the absence of disease progression or unacceptable toxicities for a maximum of 8 courses. Patients are followed every 3 months for 2 years and then at 3 years after treatment.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine and cisplatin in treating patients with metastatic breast cancer that has not responded to systemic therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate of gemcitabine and cisplatin in the treatment of metastatic breast cancer in patients who have failed one or two systemic regimens. II. Determine time to progression and survival in these patients. III. Define further the toxicity of this two-drug combination in these patients.

OUTLINE: This is a nonrandomized study. Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 1 hour on days 1, 8, and 15 every 28 days. Patients with complete response may receive an additional 2 courses after attainment of complete response status. Treatment continues in the absence of disease progression or unacceptable toxicities for a maximum of 8 courses. Patients are followed every 3 months for 2 years and then at 3 years after treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologic or cytologic confirmation of metastatic breast cancer with two exceptions: -New or enlarging pulmonary nodules demonstrable on two chest radiographs taken at least one month apart OR -Multiple characteristic lytic bone metastasis or liver metastases Measurable indicator lesion Measurable metastatic disease must be bidimensionally measurable except in the case of hepatomegaly that may be unidimensionally measurable Patients receiving bisphosphonates must have a measurable disease other than bone No CNS metastases unless controlled with prior surgery and/or radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: WBC at least 3500/mm3 or absolute neutrophil count at least 2000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 0.3 mg/dL above upper limit of normal limit (ULN) AST no greater than 3 times ULN Renal: Creatinine no greater than 0.3 mg/dL above ULN Cardiovascular: No New York Heart Association class III or IV heart disease Other: Physician-estimated oral caloric intake of at least 1200 calories per day No uncontrolled infection or chronic debilitating disease Not pregnant or nursing Women of childbearing potential must use adequate contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Must have previously received 1 but no more than 2 chemotherapy regimens At least 1 prior regimen administered for metastatic disease At least 1 prior regimen containing an anthracycline or paclitaxel At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy No prior strontium 89 radiotherapy Prior radiotherapy must have been to less than 25% of bone marrow Surgery: At least 4 weeks since any major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1997-08; Primary Completion 2005-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A. Burch, MD, Study Chair — Mayo Clinic
Locations (20):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Burch PA, Mailliard JA, Hillman DW, Perez EA, Krook JE, Rowland KM, Veeder MH, Cannon MW, Ingle JN. Phase II study of gemcitabine plus cisplatin in patients with metastatic breast cancer: a North Central Cancer Treatment Group Trial. Am J Clin Oncol. 2005 Apr;28(2):195-200. doi: 10.1097/01.coc.0000144815.54746.d0. PMID 15803016